CLINICAL TRIAL: NCT05177705
Title: The Intersection Between Loss of Control Eating and Obesity: The Role of Restriction and Food Reinforcement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Katherine Balantekin, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002806; K01DK120778 (NIH)
Record Dates: First submitted 2021-12-10; First posted 2022-01-04 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Obesity; Nutrition Disorders; Binge Eating; Body Weight
Keywords: Relative Reinforcing Value; Obesity Risk; Children; Loss of Control; Restriction
MeSH Terms: conditions — Pediatric Obesity; Nutrition Disorders; Bulimia; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Behavioral restriction (Experimental): In the restriction period participants will have their preferred (chosen after doing a preference task, including liking) food and similar alternatives restricted by their parent for 2 weeks. In the structured intake period period, participants and their parents will be given several portions of the preferred food (chosen after doing a preference task, including liking) and will consume it throughout the two-week period.
  Interventions: Behavioral: Restricted access task

INTERVENTIONS:
Behavioral: Restricted access task — In the restriction period participants will have their preferred (chosen after doing a preference task, including liking) food and similar alternatives restricted by their parent for 2 weeks. In the no restricted period, participants and their parents will be given several portions of the preferred food and will consume it throughout the two-week period.

SUMMARY:
This study aims to determine the relationships among loss of control eating, restriction, relative reinforcing value of high energy-dense food, and obesity risk. In order to achieve this aim, the investigators will follow children over the course of a year, obtaining behavioral and observational measurements, in addition to a two-week restricted access and two week non-restricted access period.

DETAILED DESCRIPTION:
The study will be mostly observational but will also include a randomized, cross-over design (the restricted access paradigm). The investigators will recruit children at risk for obesity in Erie County, New York (N=100, 50 boys, 50 girls). The study will include 4 visits at baseline and follow-up visits at 6 and 12 months. At the first visit, the participants will complete consent, height/weight/body fat, questionnaires, and complete a delayed discount task and the relative reinforcing value task. The participants will be randomized to have two weeks of restricted access first or two weeks of non-restricted access first, and then will come into the laboratory to do the loss of control test meal. Then they will have a one-week washout period, and will then complete the other two weeks of restricted/not restricted access. Following this, they will complete the loss of control test meal again. At the follow-up visits, participants will come into the laboratory to have their height/weight/body fat measured, complete questionnaires, and complete the delayed discounting task, food reinforcement and loss of control test meals. Participants will be compensated for their time after each visit. The details of the measures and procedures are outlined below.

ELIGIBILITY:
Inclusion Criteria:

* Children (male and female) ages 8-11
* At risk for obesity or with obesity (defined as either having a BMI percentile that classifies the child as having overweight-BMI >85th percentile but <99th OR one + biological parent with overweight/obesity-BMI >25)
* Rating of neutral or higher for 50% of the study foods
* Consumption of one of the study foods at least twice/week

Exclusion Criteria:

* Children below age 8 or above age 11
* Not at risk for obesity (defined as having a BMI percentile that classifies the child as having normal weight-BMI <85th percentile without having a parent with overweight or obesity)
* Allergic to study foods
* Dislike of study foods (Less than 50% of the study foods rated neutral or higher)
* Does not consume at least one study food at least twice/week
* Current diagnosis of a clinical eating disorder (ED)
* Use of medications known to affect appetite (Ritalin, Adderall, Concerta, Wellbutrin, Prednisone, etc)
* Unwillingness to complete study visits

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Change in zBMI | Baseline to 12 months
  Change in zBMI from baseline to 12 month follow-up

SECONDARY OUTCOMES:
Change in body fat percentage | Baseline to 12 months
  Change in percent body fat from baseline to 12 month follow-up
Impact of parental restriction of a High Energy Dense (HED) food on Loss of Control (LOC) eating. | Baseline
  To examine change in energy intake and macronutrient composition during LOC test meal between parental restriction condition and parental non-restriction condition.
Association between relative reinforcing value of high energy dense foods and LOC | Baseline
  Relationships will be examined between RRV and both self-reported LOC eating and intake (calories, macronutrient distribution) in the LOC test meal.
Relationship between self-reported LOC eating and consumption during LOC test meal | Baseline
  Responses between self-reported feelings of LOC and intake (calories, macronutrient distribution) will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Balantekin, PhD, RD, Principal Investigator — Clinical Associate Professor
Locations (1):
- State University of New York at Buffalo, South Campus, Buffalo, New York, United States